CLINICAL TRIAL: NCT01774201
Title: Respiratory Function and Walking Capacity in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Anna Wittrin, Phd, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OLL-260361
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Sclerosis; Respiratory; Disorder, Functional, Impaired; Difficulty Walking
Keywords: Multiple sclerosis; Self-assessment; Physical endurance; Respiratory function; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Mobility Limitation; Respiratory Aspiration; Fatigue | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breathing exercises (Experimental): Daily deep breathing exercises during two month
  Interventions: Other: Breathing exercises
- Control (No Intervention): Control group

INTERVENTIONS:
Other: Breathing exercises — Breathing exercises with positive expiratory pressure.
  Arms: Breathing exercises

SUMMARY:
Multiple sclerosis (MS) is a chronic progressive neurological disease. Respiratory dysfunction due to weakness in the respiratory musculature has been described in MS. This leads to increased morbidity and mortality in late stages of the disease. It is possible that respiratory dysfunction influence physical fitness in earlier stages as well. Walking disability and fatigue causes significant impact on health in patients with MS, even in earlier stages.

The hypothesis is that there is a relationship between respiratory function, walking capacity and fatigue and that daily deep breathing exercise during two months will improve respiratory function, walking capacity and fatigue.

DETAILED DESCRIPTION:
Presented above.

ELIGIBILITY:
Inclusion Criteria:

* Inhabitant in Orebro county, Sweden, that are diagnosed with MS according to the revised McDonald criteria and registered in the Swedish MS-registry with EDSS (Expanded disability status scale) score in the interval ≥ 3.0 - ≤ 7.0.
* Participants must understand verbal and written information and must be relapse free ≥ 3 months prior to inclusion.

Exclusion Criteria:

* Patients with diseases that may have influence on walking ability and respiratory function (other than MS). Such conditions include heart and lung diseases, orthopedic disorders, patients recently subjected to surgery, and non-MS related neurological dysfunction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | Two months
  Maximum expiratory pressure

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Westerdahl, Phd, Principal Investigator — Department of Physiotherapy, Örebro University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Westerdahl E, Wittrin A, Kanahols M, Gunnarsson M, Nilsagard Y. Deep breathing exercises with positive expiratory pressure in patients with multiple sclerosis - a randomized controlled trial. Clin Respir J. 2016 Nov;10(6):698-706. doi: 10.1111/crj.12272. Epub 2015 Mar 2. PMID 25620034
- [Result] Nilsagard Y, Westerdahl E, Wittrin A, Gunnarsson M. Walking Distance as a Predictor of Falls in People With Multiple Sclerosis. Physiother Res Int. 2016 Jun;21(2):102-8. doi: 10.1002/pri.1625. Epub 2015 Mar 17. PMID 25782023